CLINICAL TRIAL: NCT03199404
Title: TRevo Aspiration Proximal Flow Control for Endovascular Stroke Intervention Data Registry
Brief Title: Trevo Aspiration Proximal Flow Control Registry
Acronym: TRAP
Status: Terminated | Type: Observational
Why Stopped: Lead site preference
Sponsor: University of Massachusetts, Worcester (Other)
Collaborators: Stryker Neurovascular (Industry)
Responsible Party: Principal Investigator, Ajit Puri, Principal Investigator, University of Massachusetts, Worcester
Other Study IDs: TRAPv1.9
Record Dates: First submitted 2017-06-12; First posted 2017-06-26 (Actual); Last update posted 2019-10-21 (Actual); Status verified 2019-10

CONDITIONS: Stroke, Ischemic
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Treated Subjects: Subject experiencing an acute ischemic stroke in which imaging demonstrates a vascular occlusion located in the distal internal carotid artery (ICA) through the distal middle cerebral artery (MCA) and in which the TRAP technique is used for at least the first two thrombectomy passes per occluded vessel and that meet the other inclusion-exclusion criteria.
  Interventions: Device: TRAP

INTERVENTIONS:
Device: TRAP — Mechanical thrombectomy performed with the combination of a stent retriever that is partially re-sheathed and withdrawn under constant aspiration along with the use of a balloon guide catheter for distal flow control during thrombectomy.

SUMMARY:
This purpose of this retrospective, single-arm, non-randomized, multi-center study is to collect real-world data on the effectiveness of using the TRAP technique in acute ischemic stroke patients undergoing mechanical thrombectomy.

DETAILED DESCRIPTION:
The TRAP Registry is designed to collect real-world data on the use of the TRAP technique for mechanical thrombectomy in stroke patients. Recanalization success (as assessed using a TICI Score), along with the time to recanalization and number of passes needed for success will be assessed at the conclusion of the procedure. In addition, neurologic recovery (as evaluated using the Modified Rankin Scale and National Institutes of Health Score) will be assessed at 24 hours, discharge, and 90 days after the thrombectomy procedure.

ELIGIBILITY:
Inclusion Criteria:

* Subject experiencing an acute ischemic stroke in which imaging demonstrates a vascular occlusion located in the distal internal carotid artery (ICA) through the distal middle cerebral artery (MCA)
* Subjects in which the TRAP technique is used for at least the first two thrombectomy passes per occluded vessel
* Subjects that range in age from 18-85
* Subjects with a prestroke modified Rankin scale of 0-1 and presenting with an NIHSS of 8-30
* Subjects that the operator feels may be treated with endovascular therapy
* Subjects in which computed tomography (CT)/Magnetic Resonance Imaging (MRI) demonstrates an infarct size of less than 70cc on MRI or Alberta Stroke Program Early CT (ASPECTS) score overall of 6 or better
* Subjects in which groin puncture can be obtained within 6 hours of symptom onset (with or without Total Plasminogen Activator administration)
* Subjects who have consented in accordance with local Institutional Review Board requirements

Exclusion Criteria:

* Absence of large vessel occlusion on neuroimaging
* Evidence of tandem occlusion on neuroimaging
* Platelet count < 100 x 10³ cells/mm³ or known platelet dysfunction
* Contraindication to CT and/or MRI (i.e., due to contrast allergy or prior implant that precludes MRI imaging)
* Previously documented contrast allergy that is not amenable to medical treatment
* Women who are pregnant or breastfeeding at time of intervention
* Evidence of brain hemorrhage on CT and/or MRI at presenting hospital

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients presenting with acute ischemic stroke at participating hospitals in which the TRAP technique is used for mechanical thrombectomy.
Sampling Method: Non-Probability Sample
Enrollment: 38 (Actual)
Dates: Start 2017-06-06 (Actual); Primary Completion 2019-10-03 (Actual); Study Completion 2019-10-03 (Actual)

PRIMARY OUTCOMES:
Recanalization after Endovascular Intervention | Day 0: Conclusion of Thrombectomy Procedure
  Revascularization as assessed via Thrombolysis in Cerebral Infarction (TICI) score (TICI 2b/3) in affected vessels
Time to Recanalization | Day 0: Conclusion of Thrombectomy Procedure
  The time required to attain recanalization (TICI 2b/3) in affected vessels
Number of Passes for Recanalization | Day 0: Conclusion of Thrombectomy Procedure
  The total number of passes with the stent retriever need to attain recanalization will be captured.
Distal Emboli | Day 0: Conclusion of Thrombectomy Procedure
  Incidence of distal emboli (both to affected vessel and new vessel) will be assessed

SECONDARY OUTCOMES:
Neurologic Outcomes | 90 days after treatment
  Neurologic recovery as assessed by the National Institutes of Health Stroke Scale
Functional Outcomes | 90 days after treatment
  Neurologic recovery as assessed by the Modified Rankin Scale
Adverse Events | Day 1, Day 5-7 and Day 90
  Incidence of serious procedure-related adverse events will be captured
TRAP Technique | Day 0: Conclusion of thrombectomy procedure
  Success of using all components of the TRAP technique will be assessed by questionnaire for the interventionalist

CONTACTS AND LOCATIONS:
Overall Officials: Ajit Puri, MD, Principal Investigator — UMass Medical School
Locations (1):
- University of Massachusetts, Worcester, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided